CLINICAL TRIAL: NCT02998333
Title: Does Arthroscopic Anatomic Repair of the Anterior Talofibular Ligament Provide Better Functional Outcome Compared to Open Anatomic Repair in Patients With Chronic Ankle Instability: a Multicentre Randomized Controlled Trial
Brief Title: Chronic Ankle Instability, Surgical Repair: Open Versus Closed
Acronym: CAISR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gwendolyn Vuurberg (Other)
Collaborators: Zimmer Biomet (Industry); Centro Hospitalar do Porto (Other); Site Hôpital orthopédique (Unknown); Amphia Hospital (Other); Albert Schweitzer Hospital (Other)
Responsible Party: Sponsor-Investigator, Gwendolyn Vuurberg, PhD Candidate, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016_136#B2016709; NL55707.018.16 (Registry Identifier: ABR-form (toetsingonline.nl))
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Ankle Instability
Keywords: Instability; Ankle; Surgical stabilization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open surgical ankle stabilization (Active Comparator): These patients will receive open surgical stabilization of the ankle joint after failed conservative treatment with complaints for at least 6 months.
  Interventions: Procedure: Surgical stabilization
- Arthroscopic surgical ankle stabilization (Active Comparator): These patients will receive arthroscopic surgical stabilization of the ankle joint after failed conservative treatment with complaints for at least 6 months.
  Interventions: Procedure: Surgical stabilization

INTERVENTIONS:
Procedure: Surgical stabilization — Surgical stabilization of the ankle joint, performed as an open or arthroscopic procedure.

SUMMARY:
Rationale: Lateral ankle ligament injuries may be a result of ankle sprains. In 10-30% of patients with lateral ankle ligament injuries, chronic lateral ankle instability may be present. If conservative treatment fails, instability is treated surgically. Anatomic repair (also known as the Bröstrom procedure) is the current golden standard for surgical treatment of chronic ankle instability. The Bröstrom started out as an open technique and is now also performed arthroscopically. Both approaches are considered standard care and provide good results. Which approach is best, has not yet been researched. In this study it is hypothesized arthroscopic repair provides better functional outcome compared to open repair during short term follow-up.

Objective: The main objective of this study is to compare the functional outcome after arthroscopic and open anatomic repair in patients with chronic lateral ankle instability, and secondly to assess ankle stability and ankle Range of Motion (ROM) after arthroscopic and open ligament repair.

Study design: A Non-Blinded Prospective Randomized Controlled Trial Study population: All patients willing to participate, from an age of 18 years old, with persisting ankle instability for at least 6 months, eligible for anatomic repair.

Intervention: Both groups of patients are surgically treated with anatomic repair of the anterior talofibular ligament (ATFL). One group is treated arthroscopically and the other by the open approach.

Main study parameters/endpoints: The primary outcome measure is functional outcome 6 months after surgery measured using the Foot and Ankle Outcome Score. The main study parameter is a difference of ≥10 2 points per FAOS subscale between both treatment groups (Minimal Important Change = 10 points; 2 per subscale).

ELIGIBILITY:
Inclusion Criteria:

* Patients are 18 years or older;
* Experience pain and/or a sensation of instability during sports and/or daily activity;
* Isolated lateral ankle instability;
* Planned for surgical repair of the ATFL;
* At least one previous episode of an ankle inversion sprain;
* Complaints for at least 6 months;
* Failed previous conservative treatment.

Exclusion Criteria:

* Serious concomitant injury (like arthrosis, ruled out using an AP and lateral x-ray according to standard protocol);
* Foot or ankle fracture in past;
* Previous foot or ankle surgery;
* ROM restriction of >10 degrees;
* Medial instability;
* Severe misalignment;
* Ankle/foot deformities (e.g. severe flat foot);
* Systemic comorbidity leading to delayed recovery (e.g. Diabetes Mellitus, Rheumatoid Arthritis)
* (general) Hyper laxity
* Inability or unwillingness to provide consent
* Present factors that may cause difficulty of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Functional outcome | 6 months
  The primary outcome measures is a difference in pain and disability between both treatment groups as measured a Functional Ankle Outcome Score (FAOS) score change of ≥2 points per subscale measured at 6 months follow-up.

SECONDARY OUTCOMES:
Functional outcome FAOS | 3- and 6 months
  For assessment disablement
Functional outcome Numeric Rating Scale (NRS) pain | 3- and 6 months
  For pain assessment
Functional outcome Cumberland Ankle Instability Tool (CAIT) | 3- and 6 months
  For instability assessment
Anterior Drawer Test (ADT) | Pre-operative, instraoperative, 3- and 6 months postoperative
  The anterior drawer test is registered per mm (range 0-15mm) displacement and according to the manual anterior drawer test (M-ATT) categories (grade 0-3).
Range of Motion (ROM) | Pre-operative, instraoperative, 3- and 6 months postoperative
  ROM is registered in degrees of dorsi- and plantarflexion and is measured using a goniometer. Assessment is performed pre-operatively, and at 3- and 6-months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: G.M.M.J. Kerkhoffs, Professor, Principal Investigator — Department of Orthopaedic Surgery, AMC, Amsterdam, The Netherlands
Locations (3):
- AMC, Amsterdam, Netherlands
- Centro Hospitalar Povoa deVarzim, Porto, Portugal
- Site Hôpital orthopédique, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kobayashi T, Gamada K. Lateral Ankle Sprain and Chronic Ankle Instability: A Critical Review. Foot Ankle Spec. 2014 Aug 1;7(4):298-326. doi: 10.1177/1938640014539813. Epub 2014 Jun 24. PMID 24962695
- [Background] Brostrom L. Sprained ankles. VI. Surgical treatment of "chronic" ligament ruptures. Acta Chir Scand. 1966 Nov;132(5):551-65. No abstract available. PMID 5339635
- [Background] Mabit, C.C., J.M.; Fiorenza, F.; Huc, H.; Pecout, C., Lateral ligament reconstruction of the ankle: comparative study of peroneus brevis tenodesis versus periosteal ligamentoplasty. Foot and Ankle Surgery, 1998. 4(2): p. 6.
- [Background] Pereira H, Vuurberg G, Gomes N, Oliveira JM, Ripoll PL, Reis RL, Espregueira-Mendes J, Niek van Dijk C. Arthroscopic Repair of Ankle Instability With All-Soft Knotless Anchors. Arthrosc Tech. 2016 Feb 1;5(1):e99-e107. doi: 10.1016/j.eats.2015.10.010. eCollection 2016 Feb. PMID 27073785
- [Background] Drakos MC, Behrens SB, Paller D, Murphy C, DiGiovanni CW. Biomechanical Comparison of an Open vs Arthroscopic Approach for Lateral Ankle Instability. Foot Ankle Int. 2014 Aug;35(8):809-815. doi: 10.1177/1071100714535765. Epub 2014 May 21. PMID 24850160
- [Background] Matsui K, Takao M, Miyamoto W, Matsushita T. Early recovery after arthroscopic repair compared to open repair of the anterior talofibular ligament for lateral instability of the ankle. Arch Orthop Trauma Surg. 2016 Jan;136(1):93-100. doi: 10.1007/s00402-015-2342-3. Epub 2015 Oct 14. PMID 26467354